CLINICAL TRIAL: NCT00208741
Title: A 12-Week Open-Label Study Followed By A 24-Week Double-Blind Discontinuation Exploratory Study To Evaluate The Effects Of Gabitril™ (Tiagabine Hydrochloride) In Patients With Social Anxiety Disorder (SAD)
Brief Title: Study To Evaluate The Effects Of Gabitril™ In Patients With Social Anxiety Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 0337-2002
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Social Anxiety Disorder
Keywords: Social Anxiety Disorder; Mental Health
MeSH Terms: conditions — Phobia, Social; Psychological Well-Being | interventions — Tiagabine

INTERVENTIONS:
Drug: Gabitril

SUMMARY:
The main purpose of this study is to determine how safe and effective Gabitril is for outpatients with Social Anxiety Disorder (SAD).

DETAILED DESCRIPTION:
This study is being conducted at two sites in the United States. Approximately 50 patients, who are between the ages of 18 and 65 years old will be enrolled at Emory. This study consists of two parts. The first part consists of 12 weeks of open-label treatment with Gabitril. If the study doctor determines that the patients condition has improved and they have completed the initial 12 weeks of treatment they may be eligible for the second part of the study. This part is a 24-week double-blind treatment period with either Gabitril or placebo (inactive medication). There will also be a follow-up visit about 1 to 3 weeks after they have completed taking the study medication. Altogether study participation is expected to last approximately 37 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of SAD
* CGI (S) ≥ 4 at screen
* LSAS ≥ 50 at baseline
* Covi Anxiety Scale score greater than the Raskin depression Scale total score at screen

Exclusion Criteria:

* Non-responsive to adequate trials of two or more treatment medications, if previously treated for SAD.
* HAM-D ≥15 or a score of >2 on Item 1 at baseline
* Serious or unstable medical condition
* Alcohol or substance use disorder within 6 months prior to study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2002-06; Study Completion 2003-11

PRIMARY OUTCOMES:
Liebowitz Social Anxiety Scale (LSAS)
Clinical Global Impression-Change (CGI-C)

SECONDARY OUTCOMES:
Hamilton Anxiety Scale (HAM-A)
Social Phobia Inventory (SPIN)
Pittsburgh Sleep Quality Index (PSQI)
36-Item Short-Form Health Survey (SF-36)
Clinical Global Impression-S (CGI-S).

CONTACTS AND LOCATIONS:
Overall Officials: Philip T Ninan, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University School of Medicine, Atlanta, Georgia
  - Hillside Hospital of the North Shore-Long Island Jewish Health System, Long Island City, New York
  - Columbia/New York State Psychiatric Institute, New York, New York